CLINICAL TRIAL: NCT04670991
Title: Evaluation of the ExacTrac® Imaging Device for the Repositioning Quality of Patients Undergoing an External ENT Radiotherapy
Brief Title: Evaluation of ExacTrac® Imaging Device for Repositioning Quality of Patients Undergoing an External ENT Radiotherapy
Acronym: ST-IGRT-ORL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ET20-184 - ST-IGRT ORL
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Cancer; Radiotherapy Side Effect
Keywords: Cancer; Radiotherapy
MeSH Terms: conditions — Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: Monocentric, category 2 study according to Jardé Law (minimal risks and constraints) of three prospective cohorts: Tumors located at the oropharynx, the oral cavity and the larynx-hypopharynx
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXATRAC imaging (Other): For each radiotherapy session, patient will first have an Exatrac imaging and then a CBCT imaging. Patient's repositionning will be performed accoding to CBCT data
  Interventions: Radiation: EXATRAC imaging

INTERVENTIONS:
Radiation: EXATRAC imaging — Exatrac imaging performed before the standard CBCT imaging prior to each chemotherapy session

SUMMARY:
Monocentric, category 2 study according to Jardé Law (minimal risks and constraints) of three prospective cohorts: Tumors located at the oropharynx, the oral cavity and the larynx-hypopharynx.

The main objective is to evaluate the 3D vector of the absolute residual positioning error observed with the CBCT reference imaging, after repositioning performed with ExacTrac®.

The secondary objectives are to evaluate: 1) the rate of residual errors ≥2mm (translations in all directions) and ≥2 ° (rotations in all directions) on CBCT imaging after repositionning with the ExacTrac® system; 2) the Evaluation of intrafraction movements amplitude by analyzing the ExacTrac® images taken during the irradiation; 3) the evolution of the relative position of the volume of the tumor at high risk of recurrence (CTVTHR) in relation to the spine over the entire duration of the treatment; 4) the impact of patient's weight loss, the advancement of RT and the realization of a chemotherapy / targeted therapy concomitant with RT, on the evolution of the relative position of the CTVTHR in relation to the column vertebral; 5) the dosimetric consequence of a strict bone registration on the CTVTHR coverage by calculating the post-treatment dose on the CBCT imaging.

DETAILED DESCRIPTION:
The radiotherapy treatment preparation requires performing a dosimetric scanner (CT) of the patient in the treatment position, with the compression. The repositioning of the ENT sphere can be complex, especially in cases where there is irradiation of the supraclavicular lymph node areas. Indeed, the height of the irradiated area can easily exceed 20cm and it is necessary to ensure a good reproducibility of the repositioning of the spine relative to the skull.

At the end of the dosimetric CT, the radiotherapist delineates the macroscopic tumor volume (GTV) as well as the clinical tumor target volumes (CTVT) and lymph nodes (CTVN), which take into account the infiltration risks of the tissue around the macroscopic tumor. Margins around the VCTs then make it possible to obtain the estimated PTV target volumes (T and N), defined so that the VCTs receive the prescribed dose despite the geometric uncertainties associated with the treatment. Contours of organs at risk (OAR) are also carried out on the dosimetric CT. Margins around the most critical OARs (eg: marrow, brainstem, chiasma and optic nerves) are then added to generate predictive target volumes of organs at risk (PRV), taking into account the geometric uncertainties. These uncertainties are separated into errors in the treatment execution (random) and errors in the treatment preparation (systematic).

Execution errors include repositioning errors, organ movements (overnight), patient anatomical changes, intrafraction movements.

Errors related to treatment preparation include repositioning errors related to patient's skin spotting of the treatment isocenter during the dosimetric CT (thanks to room lasers), errors related to the CT acquisition that sets the CTV in a given position, the CTV delineation errors.

Dosimetry is then carried out taking into account the dose criteria to be respected on the PRVs and PTVs. Whatever the protocol used [Shrinking Action Level (SAL), non-action-level (NAL) or e-NAL (extented NAL)], it must at least make it possible to guarantee that the delivered dose complies with the planned dose. An optimization of the imaging protocol must then be able to reduce the margins without compromising the treatment quality, while reducing its toxicity for the patient.

On the Centre Léon Bérard accelerators equipped with both CBCT and ExacTrac®, we would like to assess the possibility of replacing or reducing the frequency of CBCTs using ExacTrac®. The time-consuming and irradiating characteristics of CBCT encourage to propose this study, which will define the patients for whom the use of CBCT can be minimized.

In addition, if the correlation between ExacTrac® and CBCT is good, the use of ExacTrac® will make it possible to control and correct intrafraction movements, and therefore reduce the random uncertainties associated with carrying out the treatment.

The possibility of using ExacTrac® imaging for the repositioning of patients treated with RCMI ENT would allow a reduction in treatment time and therefore less discomfort for the patient, a reduction in the dose linked to repositioning imaging, follow-up and correction of patient movements during the irradiation period.

Finally, this project will enable to propose new pre-treatment imaging strategies and personalized margins according to the position of the lesions to be treated at the ENT level in order to reduce the session time when possible, and to reduce the radiation doses. X due to imaging.

The overall objective is to improve the care and quality of treatment for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient requiring an ENT radiotherapy with intensity modulation (IMR) in the oropharynx, oral cavity, hypopharynx or larynx with bilateral irradiation of the lymph node areas
* Treatment planned on an accelerator equipped with a CBCT and the ExacTract® device
* Patient affiliated to a social security system
* Informed consent dated and signed

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient under totorship, curatorship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2024-04-13 (Estimated); Study Completion 2024-10-13 (Estimated)

PRIMARY OUTCOMES:
Verification of the feasibility of using the ExacTrac® system as a replacement for CBCT imaging for pre-treatment repositioning of ENT sphere cancers in adult patients receiving CRMI on a linear accelerator equipped with 2 modalities | Until the end of the radiotherapy treatment
  3D vector of the absolute residual positioning error observed with the CBCT reference imaging, after repositioning performed with ExacTrac®

SECONDARY OUTCOMES:
Evaluation of residual errors rates ≥2mm (translations in all directions) and ≥2 ° (rotations in all directions) on CBCT imaging after repositionning with the ExacTrac® system | Until the end of the radiotherapy treatment
  Percentage of differences in translations and rotations >2mm and 2 ° between the 2 systems
Evaluation of intrafraction movements amplitude by analyzing the ExacTrac® images taken during the irradiation | Until the end of the radiotherapy treatment
  Average of translations and rotations obtained on the intrafraction images from ExacTrac®
Evaluation of intrafraction movements amplitude by analyzing the ExacTrac® images taken during the irradiation | Until the end of the radiotherapy treatment
  Standard deviation of translations and rotations obtained on the intrafraction images from ExacTrac®
Evolution of the relative position of the volume of the tumor at high risk of recurrence (CTVTHR) in relation to the spine over the entire treatment duration | Until the end of the radiotherapy treatment
  Differential 3D vector representative of the differences in translation between a bone and a soft tissue repositionning obtained during the pre-treatment repositioning correlated with the treatment progress
Evaluation of the impact of patient's weight loss on the evolution of the relative position of the CTVTHR in relation to the spine | Until the end of the radiotherapy treatment
  Correlation between the 3D vector of absolute residual error and the evolution of the Body Mass Index
Evaluation of the impact of the RT progress on the evolution of the relative position of the CTVTHR in relation to the spine | Until the end of the radiotherapy treatment
  Correlation between the 3D vector of absolute residual error and the treatment progress
Evaluation fo the impact of a chemotherapy / targeted therapy performed concomitantly with RT, on the evolution of the relative position of the CTVTHR in relation to the spine | Until the end of the radiotherapy treatment
  Correlation between the 3D vector of absolute residual error and the administration of chemotherapy / targeted therapyconcomitantly with RT
Evaluation of the dosimetric consequence of a strict bone repositionning on the CTVTHR coverage by calculating the post-treatment dose on the CBCT imaging | Until the end of the radiotherapy treatment
  Calculation of the dose effectively delivered to target volumes and organs at risk, recalculated from pre-treatment CBCT images

CONTACTS AND LOCATIONS:
Overall Officials: BOISBOUVIER Sophie, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France